CLINICAL TRIAL: NCT00552890
Title: Influende of a Modified Atkins Diet on Glucose Metabolism and Weight Loss in Obese Type 2 Diabetic Patients - A Randomized Controlled Trial
Brief Title: Modified Atkins Diet and Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: atkins-hmo-ctil
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2001-12

CONDITIONS: Obese Type 2 Diabetic Patients
Keywords: obesity; atkins; weight reduction; kidney function
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATK (Experimental): modified Atkins diet
  Interventions: Other: modified Atkins diet
- ADA (Experimental): subjects assigned to follow ADA recommended diet for 1 year
  Interventions: Other: ADA recommended diet

INTERVENTIONS:
Other: modified Atkins diet — subjects assigned to follow modified Atkins diet for 1 year
  Arms: ATK
Other: ADA recommended diet — subjects assigned to follow ADA recommended diet for period of 1 year
  Arms: ADA

SUMMARY:
This randomized control trial compared the influence of an Atkins diet to that of the ADA recommended diet on Type 2 diabetic obese patients during a one-year follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients age 35-75 years
* BMI 30-39.9kg/m
* HbA1C>7%
* Not receiving insulin
* Micro-albumin excretion<60 mg/day

Exclusion Criteria:

* Serum creatinine level > 1.4 mg per deciliter
* Diastolic blood pressure > 100 mmHg or systolic blood pressure > 180mmHg
* Liver disease
* LDL cholesterol > 160 mg per deciliter despite lipid-lowering treatment
* Use of psychiatric medications
* Osteoporosis
* Cancer
* Food allergies, and
* Low carbohydrate diet in the past 6 months.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2001-12; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
weight loss and glucose control | 1 year

SECONDARY OUTCOMES:
lipid profile, kidney function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Director, Diabetes Unit, Hadassah University Hospital